CLINICAL TRIAL: NCT04912752
Title: Copy Number Variation in Migraine and Gene Expression
Brief Title: Copy Number Variation in CHRNA7 Gene in Migraine and Gene Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Şenay Görücü Yılmaz, Assoc. Prof., University of Gaziantep
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2020/12
Record Dates: First submitted 2021-05-21; First posted 2021-06-03 (Actual); Last update posted 2021-06-03 (Actual); Status verified 2021-05

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case-Control (Other): Copy number variation
  Interventions: Genetic: Migraine CNV
- Case-Control 1 (Experimental): Gene expression
  Interventions: Genetic: Migraine CNV

INTERVENTIONS:
Genetic: Migraine CNV — Copy number variation effect on migraine disease

SUMMARY:
Migraine is a common and possible hereditary disease. Copy number variation (CNV) is a phenomenon in which parts of the genome are repeated and the number of repeats in the genome varies between individuals in the human population.The CHRNA7 gene has a major role in the neuropsychiatric phenotypes observed in patients. The 15q13.3 gain/loss variation in this gene may be associated with migraine.

DETAILED DESCRIPTION:
Migraine is a common neurological disorder. Although they have different genetic bases according to their types, cholinergic receptors after calcium channels play an important role in the clinic and genetics of the disease. Neuronal acetylcholine receptor subunit alpha-7, also known as nAChRα7, is a protein that in humans is encoded by the CHRNA7 gene.

ELIGIBILITY:
Inclusion Criteria:

Migraine

Exclusion Criteria:

Vascular problems

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-04-05 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-01-02 (Actual)

PRIMARY OUTCOMES:
CNV number | 1 year
  CNV number effect on migraine

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Fatih Özaltun, MD, Principal Investigator — Assist
Locations (1):
- Medicine, Gaziantep, Şehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
manuscript not yet published